CLINICAL TRIAL: NCT03113851
Title: Observation of Abscopal Effect of Radiation in Combination With rhGM-CSF for Patients With Metastatic Non-small Cell Lung Cancer
Brief Title: Abscopal Effect of Radiation in Combination With rhGM-CSF for Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Anhui Shi, MD, Associate Chief Physician, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016YJZ23
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer Metastatic
MeSH Terms: interventions — Radiotherapy; Radiation; regramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy and rhGM-CSF (Experimental): Patients with metastatic non-small cell lung cancer received 3.5 Gy per fraction to a total dose of 35 Gy/ 10 fractions over 2 weeks, combined with rhGM-CSF (125 μg/m2).
  Interventions: Radiation: Radiotherapy; Drug: rhGM-CSF

INTERVENTIONS:
Radiation: Radiotherapy — One lesion received radiotherapy for 35 Gy in 10 fractions and rested for one week; then another metastatic lesion were treated with radiotherapy for 35 Gy in 10 fractions.
  Other Names: radiation
Drug: rhGM-CSF — Patients were injected subcutaneously rhGM-CSF 125mg/m2 per day from day1 to day 14, every three weeks, concurrent with radiotherapy
  Other Names: recombinant human GM-CSF

SUMMARY:
The purpose of this study is to determine whether radiation combined with recombined human granulocyte-macrophage colony stimulating factor(rhGM-CSF) is safe and effective for patients with metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
The prognosis of patients with metastatic non-small cell lung cancer was still poor for those unsuitable for target therapy or immunotherapy. This study is to include patients evaluated as effective or stable disease after first-line chemotherapy or progressed after second-line chemotherapy to evaluate the efficacy and safety of receiving radiotherapy combined with recombined human granulocyte-macrophage colony stimulating factor(rhGM-CSF).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histologically proven non-small-cell lung cancer；
3. Stage IV according to UICC stage system(version 7,2009), at least with three evaluable abscopal lesions (≥1cm)（excluding intestinal metastasis）;
4. Evaluated as effective or stable disease after first-line chemotherapy or progressed after second-line chemotherapy (progression sites were no more than three sites);
5. ECOG performance status: 0-1;
6. Life expectancy ≥ 3 months.
7. Adequate baseline organ and marrow function: absolute neutrophil count greater than 1500 cells per μL, platelet concentration of greater than 50 000 per μL, total bilirubin less than 1•5 times the upper limit of normal (ULN), aspartate aminotransferase and alanine aminotransferase less than 2•5 times the ULN, and serum creatinine less than 1•5 times the ULN;
8. Female subjects have a negative urine or serum pregnancy test within 1 week prior to treatment if of childbearing potential;
9. Asymptomatic subjects with brain metastasis can be included, but the sites of brain cannot be considered as target sites;
10. Asymptomatic subjects with bone metastasis can be included, but the sites of bone cannot be considered as target sites.

Exclusion Criteria:

1. Having received immunotherapy within 4 weeks prior to inclusion;
2. Allergic to GM-CSF, or diagnosed with immune system disease, receiving immunosuppressant, such as prednisone, dexamethasone, methylprednisolone, methotrexate, hydroxychloroquine, cyclophosphamide, azathioprine and so one;
3. receiving treatment of other trials;
4. Any unstable systemic disease, including active infection, symptomatic congestive heart failure, myocardial infarction onset six months before included into the group, unstable angina, and severe arrhythmia, uncontrolled chronic lung disease;
5. unwilling to sign consent;
6. Women in pregnancy or lactation;
7. Other malignancy except for non-melanoma carcinoma of the skin or in situ carcinoma of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
The abscopal effect rate | up to 50 months
  The proportion of patients with an abscopal response assessed after the initiation of treatment

SECONDARY OUTCOMES:
Progression free survival | up to 84 months
  From the date of enrollment to the date of progression or death
Overall survival | up to 84 months
  From the date of enrollment to the date of death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anhui Shi, MD., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided